CLINICAL TRIAL: NCT03668925
Title: Association Between Hidradenitis Suppurativa and Spondyloarthritis
Acronym: VESPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PJ12076
Record Dates: First submitted 2018-08-07; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Hidradenitis Suppurativa
Keywords: spondyloarthritis; hidrosadenitis suppurativa; inflammation; magnetic resonance imaging
MeSH Terms: conditions — Hidradenitis Suppurativa; Spondylarthritis; Inflammation | interventions — Magnetic Resonance Spectroscopy; Weights and Measures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "Case" (Experimental): patient diagnosed with hidrosadenitis suppurativa
  Interventions: Radiation: magnetic resonance imaging (MRI) of the sacro-iliac region HLA B27 test C-reactive protein (CRP) measurement
- Group "control" (Active Comparator): patient without hidrosadenitis suppurativa
  Interventions: Radiation: magnetic resonance imaging (MRI) of the sacro-iliac region HLA B27 test C-reactive protein (CRP) measurement

INTERVENTIONS:
Radiation: magnetic resonance imaging (MRI) of the sacro-iliac region HLA B27 test C-reactive protein (CRP) measurement — magnetic resonance imaging (MRI) of the sacro-iliac region HLA B27 test C-reactive protein (CRP) measurement

SUMMARY:
Hidradenitis suppurativa is a chronic dermatosis, characterized by an inflammation of the follicular epithelium in the apocrine glands.

The hypothesis of a link between hidradenitis suppurativa and inflammatory rheumatism has been widely considered, with evidence in support of this theory accumulating from several case reports and small series. The most frequently cited rheumatismal disease thought to be associated with Hidradenitis suppurativa is spondyloarthritis.

Taken together, these data suggest that there may a link between hidradenitis suppurativa and spondyloarthritis, but literature data are sparse, and to date, no study has investigated or demonstrated such a relation. Indeed, existing studies to date were observational, descriptive, and retrospective, and did not use modern diagnostic approaches for documenting spondyloarthritis, such as magnetic resonance imaging (MRI) or the recent classification of spondyloarthritis.

DETAILED DESCRIPTION:
The aim of the study was to test the hypothesis that the risk of spondyloarthritis is increased in patients with hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* for case: patients with diagnosis of hidrosadenitis suppurativa in the Department of Dermatology of the University Hospital of Reims, regardless of the stage of severity and duration of their disease
* for control: patients without diagnosis of hidrosadenitis suppurativa matched to cases for age (±5 years) and sex
* for case and control: have accepted to take part in the research

Exclusion Criteria:

* for case and control: age <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
spondyloarthritis | Day 0
  spondyloarthritis was diagnosed by a rheumatologist using the Assessment of SpondyloArthritis international Society (ASAS) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Fauconier M, Reguiai Z, Barbe C, Colosio A, Eschard JP, Salmon JH, Direz G. Association between hidradenitis suppurativa and spondyloarthritis. Joint Bone Spine. 2018 Oct;85(5):593-597. doi: 10.1016/j.jbspin.2017.09.005. Epub 2017 Sep 28. PMID 28965938